CLINICAL TRIAL: NCT03812705
Title: Fecal Microbiota Transplantation for the Treatment of Steroid Resistant/Dependent Acute Gastrointestinal Graft Versus Host Disease
Brief Title: Fecal Microbiota Transplantation for Steroid Resistant/Dependent Acute GI GVHD
Acronym: FEMITGIGVHD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Liping Wan, Chief physician, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHSYXY-FMT-GVHD-2018002
Record Dates: First submitted 2019-01-19; First posted 2019-01-23 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm
Keywords: allogeneic hematopoeitic stem cell transplantation; acute gastrointestinal graft versus host disease; fecal microbiome transplantation
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Intervention Model Description: fecal microbiome transplantation for patients with steroid resistant/dependent acute gastroinstestinal graft versus host disease
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- fecal microbiome transplantation (Experimental): 1. Perform fecal microbiome transplantation to patient under colonoscopy or gastroscopy: injection of 200~300 ml fecal microbiome fluid as fecal microbiome transplantation to left colon by Colonoscopy or duodenum through duodenum tube by gastroscopy;
  2. If patient's condition is stable or improved within 1 week, second fecal microbiome transplantation may be performed 1 week later, up to 4 times will be performed if patient response;
  3. If patient's condition is not improved after the second fecal microbiome transplantation, stop fecal microbiome transplantation.
  Interventions: Biological: fecal microbiome transplantation

INTERVENTIONS:
Biological: fecal microbiome transplantation — 1. Stop antibiotics treatment 1 day before fecal microbiome transplantation;
  2. Fasting food 6 hours before fecal microbiome transplantation;
  3. Give Ondansetron intravenously 1 hour before fecal microbiome transplantation for vomiting prevention;
  4. Perform fecal microbiome transplantation under colonoscopy or gastroscopy;
  5. Perform up to 4 times if patient response;
  6. Stop if no response after twice fecal microbiome transplantation.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of fecal microbiome transplantation in patients with steroid resistant/dependent acute gastrointestinal graft-versus-host disease (GVHD). The patient will cease antibiotics treatment 1 day before FMT, and stop taking food 6 hours before FMT. Patients will be given Ondansetron intravenously 1 hour before FMT. Patients will be injected 200~300 ml fecal microbiome fluid to left colon by Colonoscopy or duodenum through duodenal tube by gastroscopy. If patient's condition is stable or improved within 1 week, second FMT may be performed 1 week later, up to 4 times will be performed if patient response. If patient's condition is not improved after the second FMT, ceasing FMT.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the efficacy and safety of fecal microbiome transplantation in patients with steroid resistant/dependent acute gastrointestinal graft-versus-host disease (GVHD).

Inclusion criteria:

1. Age>= 14 yrs ≤60 yrs.
2. Diagnosed with hematological diseases.
3. Recipients of allogeneic peripheral blood stem cell transplantation.
4. Steroid resistant/dependent acute intestinal graft-versus-host disease (GVHD) within 100 days post-transplantation. The definition of steroid resistant/dependent acute intestinal GVHD is progression within 3 days of starting treatment or an incomplete response by 7 days or recurrence after initial dose reduction.
5. ECOG score ≤2;
6. signed consent form.

Exclusion criteria:

1. Complicated with uncontrolled severe infection except intestine and colon.
2. High risk of hemorrhage, dysfunction of coagulation, active gastrointestinal hemorrhage;
3. Absolute neutrophil count (ANC) <0.5×10e9/L or platelet count (PLT) < 20×10e9/L
4. Severe organ dysfunction, including heart failure, respiratory failure, renal failure, epilepsy or central nervous system dysfunction.
5. Participating other clinical trials.
6. Pregnant women.

Treatment:

1. Stop antibiotics treatment 1 day before FMT;
2. Fasting food 6 hours before FMT;
3. Give Ondansetron intravenously 1 hour before FMT for vomiting prevention;
4. Injection of 200~300 ml fecal microbiome fluid to left colon by Colonoscopy or duodenum through duodenum tube by gastroscopy;
5. If patient's condition is stable or improved within 1 week, second FMT may be performed 1 week later, up to 4 times will be performed if patient response;
6. If patient's condition is not improved after the second FMT, stop FMT.

Major endpoint Response rate of acute gastrointestinal GVHD with 12 weeks after FMT, including complete response and partial response.

Minor endpoints:

1. Time to response of acute gastrointestinal GVHD;
2. Duration of response of acute gastrointestinal GVHD.

ELIGIBILITY:
Inclusion Criteria:

1. Age>= 14 yrs ≤60 yrs.
2. Diagnosed with hematological diseases.
3. Recipients of allogeneic peripheral blood stem cell transplantation.
4. Steroid resistant/dependent acute intestinal graft-versus-host disease (GVHD) within 100 days post-transplantation. The definition of steroid resistant/dependent acute intestinal GVHD is progression within 3 days of starting treatment or an incomplete response by 7 days or recurrence after initial dose reduction.
5. Eastern Cooperative Oncology Group (ECOG) score ≤2;
6. Signed consent form.

Exclusion Criteria:

1. Complicated with uncontrolled severe infection except intestine and colon.
2. High risk of hemorrhage, dysfunction of coagulation, active gastrointestinal hemorrhage;
3. Absolute neutrophil count (ANC) <0.5×10e9/L or platelet count (PLT) < 20×10e9/L
4. Severe organ dysfunction, including heart failure, respiratory failure, renal failure, epilepsy or central nervous system dysfunction.
5. Participating other clinical trials.
6. Pregnant women.

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2018-12-13 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Response rate | 12 weeks within FMT
  Response rate of acute gastrointestinal GVHD after FMT, including complete response and partial response.

SECONDARY OUTCOMES:
Time to response | 12 weeks within FMT
  Time to response of acute gastrointestinal GVHD
Duration of response | 12 weeks within FMT
  Duration of response of acute gastrointestinal GVHD

CONTACTS AND LOCATIONS:
Overall Officials: Liping Wan, MD, Principal Investigator — Shanghai Jiao Tong University Affiliated Shanghai General Hospiatal
Locations (2):
- China (2):
  - Shanghai Jiao Tong University Affilated First People's Hospital, Shanghai, Shanghai Municipality
  - Shanghai Jiao Tong University Affilated Shanghai General Hospital, Shanghai, Shanghai Municipality